CLINICAL TRIAL: NCT01654497
Title: A Phase I, Sequential Cohort, Open-Label, Dose-escalation Study of the Safety and CNS Pharmacokinetics of Dexanabinol in Patients With Brain Cancer
Brief Title: Dexanabinol in Patients With Brain Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santosh Kesari, M.D., Ph.D. (Other)
Collaborators: e-Therapeutics PLC (Industry)
Responsible Party: Sponsor-Investigator, Santosh Kesari, M.D., Ph.D., Associate Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111827
Record Dates: First submitted 2012-07-16; First posted 2012-07-31 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Brain Cancer
Keywords: Brain; Glioma; glioblastoma; metastases; cancer; ETS2101; leptomeningeal; astrocytoma; oligodendroglioma; meningioma
MeSH Terms: conditions — Brain Neoplasms; Glioma; Glioblastoma; Neoplasm Metastasis; Neoplasms; Astrocytoma; Oligodendroglioma; Meningioma | interventions — HU 211

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dexanabinol (Experimental)
  Interventions: Drug: Dexanabinol

INTERVENTIONS:
Drug: Dexanabinol — Dexanabinol: intravenous infusion over 3 hours, weekly (i.e., Day 1, 8, 15 and 22 of a 28-day cycle)
  Nine dosing cohorts are planned, with the option to enroll additional cohorts based on safety and PK data.
  Dose Level 1: 2 mg/kg
  Dose Level 2: 4 mg/kg
  Dose Level 3: 8 mg/kg
  Dose Level 4: 16 mg/kg
  Dose Level 5: 24 mg/kg
  Dose Level 6: 28 mg/kg
  Dose Level 7: 36 mg/kg
  Dose Level 8: 40 mg/kg
  Dose Level 9: 44 mg/kg

SUMMARY:
The purpose of this study is to try to determine the maximum safe dose of dexanabinol that can be administered to people with brain cancer. Other purposes of this study are to:

* find out what effects (good and bad) dexanabinol has;
* see how much drug gets into the body by collecting blood and cerebrospinal fluid for use in pharmacokinetic (PK) studies;
* learn more about how dexanabinol might affect the growth of cancer cells;
* look at biomarkers (biochemical features that can be used to measure the progress of disease or the effects of a drug).

DETAILED DESCRIPTION:
Protection from apoptosis is a key survival factor for cancer cells. Dexanabinol is under investigation as a novel anti-cancer therapy based on its tumoricidal activity observed in vitro and in vivo, presumably due to inhibitory activity against NFĸB, TNFα, COX-2 and additional putative targets suck as HAT, FAT and cyclin dependent kinases. Targeted induction of apoptosis in cancer cells versus normal cells provides an attractive strategy for the treatment of brain cancer, a pernicious disease with debilitating neurological side effects and poor prognoses. A single intravenous dosing of dexanabinol has demonstrated safety in humans. Therefore, we are conducting a phase I dose escalation study to examine the safety of multiple dosing of dexanabinol and drug penetration into the brain, and to determine a suitable dose for moving into a phase II trial for efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or radiologically confirmed diagnosis of brain cancer:

  * glioblastoma (GBM),
  * anaplastic astrocytoma (AA),
  * anaplastic oligodendroglioma (AO),
  * anaplastic mixed oligoastrocytoma (AMO),
  * low grade gliomas,
  * brain metastases,
  * meningiomas, or
  * leptomeningeal metastases
* Has failed prior standard therapy including maximal safe surgical resection, radiation therapy (when appropriate for the specific cancer type), and systemic therapy.
* For diagnosis of GBM: has undergone at least one prior surgical gross-total or subtotal tumor resection, a course of postoperative radiation therapy with concurrent temozolomide, and at least 2 cycles of maintenance temozolomide.
* For diagnosis of meningioma: has no other option of standard therapy such as surgical resection (partial or total resection) or radiation.
* Has progression of brain cancer and measurable disease by magnetic resonance imaging (MRI) or computed tomography (CT) scan.
* Age ≥ 18 years.
* Karnofsky Performance Status ≥ 60%. (Appendix A). Subjects must have a life expectancy of equal to or greater than 8 weeks.
* Organ and Marrow Function Requirements

Hematology:

* Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
* Platelet count ≥ 100 x 109/L
* Hemoglobin ≥ 9.0 g/dL
* White blood cell (WBC) count ≥ 3.0 x 109/L

Biochemistry:

* AST/SGOT and ALT/SGPT ≤ 2.5 x institution's ULN
* Total bilirubin ≤ 1.5 x institution's ULN
* Serum creatinine ≤ 1.5 x institution's ULN or 24-hour creatinine clearance ≥ 50 ml/min
* Alkaline phosphatase (ALP) ≤ 2.5 x ULN unless considered tumor related
* Estimated GFR > 50 ml/min (based on Wright formula)

Coagulation:

* INR < 1.5 x institution's ULN
* PT/aPTT within institution's normal range, unless receiving therapeutic low molecular weight heparin

  * Contraception Woman of child-bearing potential and man with partners of child-bearing potential agrees to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days following completion of therapy.
  * Woman of child-bearing potential has negative pregnancy test before the initiation of study drug dosing.

Exclusion Criteria:

* Current or anticipated use of other investigational agents.
* Current or anticipated use of enzyme-inducing anti-epileptic drugs (EIAED).
* Insufficient time for recovery from prior therapy:

  * less than 28 days from any investigational agent,
  * less than 28 days from prior cytotoxic therapy (except 23 days from prior temozolomide, 14 days from vincristine, 42 days from nitrosoureas, 21 days from procarbazine administration), and
  * less than 7 days for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count).
* Less than 4 weeks from surgery or insufficient recovery from surgical-related trauma or wound healing.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dexanabinol.
* History of allergic reactions to medicines containing polyoxyethylated castor oil that are not controlled with premedications.
* Severe or uncontrolled medical disorder that would, in the investigator's opinion, impair ability to receive study treatment (i.e., uncontrolled diabetes, chronic renal disease, chronic pulmonary disease or active, uncontrolled infection).
* Electrolyte abnormality that cannot be corrected to normal levels prior to initiating study drug.
* Known diagnosis of human immunodeficiency virus (HIV) infection.
* Impaired cardiac function including any of the following:

  * Congenital long QT syndrome or a known family history of long QT syndrome;
  * History or presence of clinically significant ventricular or atrial tachyarrhythmias
  * Clinically significant resting bradycardia (< 50 beats per minute)
  * Inability to monitor the QT interval by ECG
  * QTc > 450 msec on baseline ECG. If QTc > 450 and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc
  * Myocardial infarction within 1 year of starting study drug
  * Other clinically significant heart disease (e.g., unstable angina, congestive heart failure, or uncontrolled hypertension)
* Pregnant or nursing. There is a potential for congenital abnormalities and for this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-06; Primary Completion 2015-09 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities and the maximum tolerated dose (MTD) of weekly dexanabinol | first 28 days of treatment

SECONDARY OUTCOMES:
Treatment-emergent adverse events | 7 months
  description, timing, grade [CTCAE v4.03], severity, seriousness, and relatedness
Objective response rate and best overall response rate over time as assessed by the RANO criteria | approximately 6 months to 1 year
Progression free survival | up to 5 years
Overall Survival | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Santosh Kesari, MD, PhD, Principal Investigator — University of California Medical Center
Locations (1):
- Moores UCSD Cancer Center, La Jolla, California, United States